CLINICAL TRIAL: NCT04176341
Title: Feasibility and Clinical Impact Study of Non Pharmacological Interventions Targeting the Subject's Empowerment Among Slackline, Mindfulness, Adapted Physical Activity, Self-hypnosis, Qi Gong Versus Usual Care in Management of Chronic Pain
Brief Title: Feasability and Clinical Impact Study of Non Pharmacological Interventions in Management of Chronic Pain
Acronym: ELISAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Hospices Civils de Lyon (Other); Groupe Hospitalier Mutualiste de Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC19.143
Record Dates: First submitted 2019-11-15; First posted 2019-11-25 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2021-09

CONDITIONS: Chronic Pain; Slackline; Mindfulness; Adapted Physical Activity; Self-hypnosis; Qi Gong
Keywords: non pharmacological interventions; chronic pain; slackline; mindfulness; adapted physical activity; self-hypnosis; Qi Gong; shared decision making
MeSH Terms: conditions — Chronic Pain | interventions — Mindfulness; Hypnosis; Qigong

STUDY DESIGN:
Intervention Model Description: Intervention group : chronic pain patient consulting in Grenoble Alps University Hospital and Grenoble Hospital Mutualist Group who will one non pharmacological intervention between slackline, mindfulness, adapted physical activity, self-hypnosis, Qi Gong during 6 to 8 weeks.
  Control group : chronic pain patient consulting in Lyon University Hospital who will receive usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): chronic pain patient consulting in Grenoble Alps University Hospital, and Hospital Mutualist Group who will one non pharmacological intervention between slackline, mindfulness, adapted physical activity, self-hypnosis, Qi Gong during 6 to 8 weeks.
  Interventions: Other: a systematic proposal for non pharmacological interventions targeting the subject's empowerment among slackline, mindfulness, adapted physical activity, self-hypnosis, and Qi Gong
- Control group (No Intervention): chronic pain patient consulting in Lyon University Hospital who will receive usual care.

INTERVENTIONS:
Other: a systematic proposal for non pharmacological interventions targeting the subject's empowerment among slackline, mindfulness, adapted physical activity, self-hypnosis, and Qi Gong — chronic pain patient consulting in Grenoble Alps University Hospital, and Hospital Mutualist Group who will one non pharmacological intervention between slackline, mindfulness, adapted physical activity, self-hypnosis, Qi Gong during 6 to 8 weeks.
  Other Names: non pharmacological interventions
  Arms: Intervention group

SUMMARY:
This feasability study aims to compare the 6-month success rate of a systematic proposal for non pharmacological interventions targeting the subject's empowerment among slackline, mindfulness, adapted physical activity, self-hypnosis, and Qi Gong versus usual care in the management of chronic pain.

DETAILED DESCRIPTION:
Chronic pain management is complex. 27.2 to 43.5 % of general population suffers from it. Opoid crisis has shown the limit of the WHO 3 step analgesic ladder. Multidisciplinary pain management programs, shared decision making and non pharmacological interventions targeting subject's empowerment are needed. Among these non pharmacological interventions, patients are increasingly turning to traditional and complementary medicines. Evidence about their safety and efficacy is hard to build. Thus our study aims to assess the feasibility of a systematic proposal for non pharmacological interventions targeting the subject's empowerment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stable chronic pain defined by the presence of pain for more than 3 months and without substantial change in management in the month prior to inclusion
* Patient with a mean EVA maximum daily pain over 7 days greater than or equal to 4/10
* Patient aged 18 and over
* Informed and written consent signed by the patient (or his / her legal representative).
* Person affiliated with social security or beneficiary of such a scheme

Exclusion Criteria:

* Patient with a cluster headache
* Patient followed for 7 years or more by a pain center
* Patient treated with adjuvant or neo-adjuvant chemotherapy or radiotherapy for the primary tumor
* Patient with a decompensated psychiatric condition
* Patient currently participating or having participated in the month prior to inclusion in another interventional clinical research that may impact the study; this impact is left to the investigator's discretion
* Protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Compare the 6-month success rate of a systematic proposal for non pharmacological interventions targeting the subject's empowerment versus usual care in the management of chronic pain | 6 months
  The success of the intervention will be defined as a reduction of 30% or more of the average daily Visual Analog Score [0-10] for pain collected the 7 days prior to the M6 visit, compared to baseline status before intervention.

SECONDARY OUTCOMES:
Compare the effectiveness of the intervention versus usual care between M6-M3-M0 | 3 and 6 months
  Average daily pain visual analogue scale collected the 7 days prior to the visit of M0, M3 and M6.
  We will perform a subgroup analysis per workshop if n ≥ 25 in this one.
Describe adherence of the intervention | 6 months
  Number of participated workshops by patients
Describe side effects of the intervention | 6 months
  Report eventuels side effects occuring during interventions
Compare changes in quality of life at 3 and 6 months compared to baseline. | 3 and 6 months
  Evolution of the generic quality of life measured by the EQ5D-3L questionnaire at 3 and 6 months compared to baseline
Evaluate the evolution of the overall motivation of the subjects of the Intervention group at different times of the study: before, during, just after the intervention, and at 3 and 6 months. | 3 and 6 months
  Evaluate the evolution of the overall motivation (EMG-28 scale) at 3 and 6 months compared to baseline for the subjects of the Intervention group.
  To evaluate the motivation of the subjects of the intervention group with Likert scales (importance / confidence / disposition) before, during, just after the intervention, and at 3 and 6 months.
Evaluate the evolution of the detailed motivation of the subjects of the Intervention group at different times of the study: before, during, just after the intervention, and at 3 and 6 months. | 3 and 6 months
  Evaluate motivation of the subjects of the intervention group with Likert scales (importance / confidence / disposition) before, during, just after the intervention, and at 3 and 6 months.
Compare the evolution of the health care consumption of the subjects at 3 and 6 months compared to baseline. | 3 and 6 months
  Count drug consumption, herbal medicine, homeopathy, food supplements, use of care (medical consultations, hospitalization, use of complementary medicines (acupuncture, osteopathy, micro physiotherapy, chiropractic ...), professional absenteeis that occurs to patient during the study.
Evaluate the success of the intervention (intervention group) or the conventional follow-up (control group) from the patient's point of view at 3 and 6 months compared to baseline. | 3 and 6 months
  Binary success / failure criterion chosen by the patient during the inclusion visit among 5 criteria previously defined by a focus group of chronic pain patients upstream of the study, at 3 and 6 months compared to baseline.
Sub-group analysis for healthcare professionals : compare the 6-month success rate of a systematic proposal for non pharmacological interventions targeting the subject's empowerment versus usual care in the management of chronic pain | 6 months
  Sub-group analysis for healthcare professionals of the success of the intervention defined as a reduction of 30% or more of the average daily Visual Analog Score [0-10] for pain collected the 7 days prior to the M6 visit, compared to baseline status before intervention.
Compare the evolution of the ability to cope with subjects at 3 and 6 months compared to baseline. | 3 and 6 months
  Evolution of the Ways of Coping Checklist on the patient's ability to cope at 3 and 6 months compared to baseline
Compare the evolution of the catastrophism of the subjects at 3 and 6 months compared to baseline. | 3 and 6 months
  Evolution of the PCS-CF Pain Catastrophism Scale [0-52] at 3 and 6 Months compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Maindet, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU de GRENOBLE ALPES, Grenoble, France

REFERENCES:
- [Background] Shipton EA, Shipton EE, Shipton AJ. A Review of the Opioid Epidemic: What Do We Do About It? Pain Ther. 2018 Jun;7(1):23-36. doi: 10.1007/s40122-018-0096-7. Epub 2018 Apr 6. PMID 29623667
- [Background] Skelly AC, Chou R, Dettori JR, Turner JA, Friedly JL, Rundell SD, Fu R, Brodt ED, Wasson N, Winter C, Ferguson AJR. Noninvasive Nonpharmacological Treatment for Chronic Pain: A Systematic Review [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2018 Jun. Report No.: 18-EHC013-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK519953/ PMID 30179389
- [Background] Devan H, Hale L, Hempel D, Saipe B, Perry MA. What Works and Does Not Work in a Self-Management Intervention for People With Chronic Pain? Qualitative Systematic Review and Meta-Synthesis. Phys Ther. 2018 May 1;98(5):381-397. doi: 10.1093/ptj/pzy029. PMID 29669089
- [Background] Dworkin RH, Turk DC, McDermott MP, Peirce-Sandner S, Burke LB, Cowan P, Farrar JT, Hertz S, Raja SN, Rappaport BA, Rauschkolb C, Sampaio C. Interpreting the clinical importance of group differences in chronic pain clinical trials: IMMPACT recommendations. Pain. 2009 Dec;146(3):238-244. doi: 10.1016/j.pain.2009.08.019. PMID 19836888
- [Background] Olsen MF, Bjerre E, Hansen MD, Tendal B, Hilden J, Hrobjartsson A. Minimum clinically important differences in chronic pain vary considerably by baseline pain and methodological factors: systematic review of empirical studies. J Clin Epidemiol. 2018 Sep;101:87-106.e2. doi: 10.1016/j.jclinepi.2018.05.007. Epub 2018 May 21. PMID 29793007